CLINICAL TRIAL: NCT00562484
Title: A Phase IV, Randomized, Observer-Blind, Placebo-Controlled, Multi-Centre Study to Evaluate the Efficacy, Safety and Tolerability of CSL Limited's Influenza Virus Vaccine in Adults Aged ≥ 18 to < 65 Years.
Brief Title: A Study of the Efficacy, Safety and Tolerability Profile of CSL Limited's Influenza Virus Vaccine (CSL's IVV) Administered Intramuscularly in Healthy Adults
Acronym: CSL's IVV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CSLCT-USF-06-28
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Results first posted 2011-09-12 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: CSL Limited Influenza Vaccine
- 2 (Other)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CSL Limited Influenza Vaccine — A single 0.5 mL, intramuscular Injection in the deltoid region of the arm on day 0.
  Arms: 1
Biological: Placebo — Placebo
  Arms: 2

SUMMARY:
This study will assess the Efficacy, Safety and Tolerability profile of CSL's Influenza Vaccine administered intramuscularly against laboratory-confirmed influenza illness in a population defined as being not at risk of severe complications following influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged ≥ 18 to < 65 years at the time of vaccination
* Non pregnant/ non lactating females

Exclusion Criteria:

* Hypersensitivity to influenza vaccine or allergy to any components of the Study Vaccines
* Vaccination against influenza in the previous 6 months
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality
* Known history of Guillain-Barré Syndrome;
* Clinical signs of active infection and/or an oral temperature of ≥ 37.8 oC.
* History of neurological disorders or seizures
* Confirmed or suspected immunosuppressive condition or a previously diagnosed immunodeficiency disorder
* Current or recent immunosuppressive or immunomodulative therapy, including systemic corticosteroids
* Administration of immunoglobulins and/or any blood products;
* Participation in a clinical trial or use of an investigational compound;
* Vaccination with a registered vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior;
* Participants indicated to receive an influenza vaccine on an annual basis according to the local public health recommendations.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7500 (Actual)
Dates: Start 2008-03; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Vaccines, Study Director — Seqirus
Locations (24):
- Australia (20):
  - The Clinical Trials Unit, Canberra Hospital, Canberra, Australian Capital Territory
  - Australian Clinical Research Organisation, Brookvale, New South Wales
  - Australian Clinical Research Organisation, Caringbah, New South Wales
  - Eastern Area Health Service, Prince of Wales Hospital, Randwick, New South Wales
  - National Centre for Immunisation Research & Surveillance (NCIRS) The Children's Hospital at Westmead, Westmead, New South Wales
  - Australian Clinical Research Organisation, Auchenflower, Queensland
  - Trialworks Clinical Research Services, Brisbane, Queensland
  - Australian Clinical Research Organisation Caboolture Clinical Research Centre, Caboolture, Queensland
  - School of Medicine, James Cook University, Cairns Base Hospital, Cairns, Queensland
  - Gold Coast Hospital, Gold Coast, Queensland
  - Australian Clinical Research Organisation, Kippa-Ring, Queensland
  - CMAX, a division of IDT Australia, Adelaide, South Australia
  - Paediatric Trials Unit, Women's and Children's Hospital, Adelaide, South Australia
  - Primary Old Port Road Medical and Dental Centre, Royal Park, South Australia
  - Sexual Health Service, Hobart, Tasmania
  - Barwon Health, Geelong Hospital, Geelong, Victoria
  - Emeritus Research, Malvern East, Victoria
  - Murdoch Childrens Research Institute, Melbourne, Victoria
  - Lung Institute of Western Australia, Perth, Western Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- New Zealand (4):
  - Auckland Clinical Studies, Auckland
  - 198 Youth Health Centre, Christchurch
  - Southern Clinical Trials, Christchurch
  - RMC Medical Centre, Dunedin

REFERENCES:
- [Derived] Mcbride WJH, Abhayaratna WP, Barr I, Booy R, Carapetis J, Carson S, De Looze F, Ellis-Pegler R, Heron L, Karrasch J, Marshall H, Mcvernon J, Nolan T, Rawlinson W, Reid J, Richmond P, Shakib S, Basser RL, Hartel GF, Lai MH, Rockman S, Greenberg ME. Efficacy of a trivalent influenza vaccine against seasonal strains and against 2009 pandemic H1N1: A randomized, placebo-controlled trial. Vaccine. 2016 Sep 22;34(41):4991-4997. doi: 10.1016/j.vaccine.2016.08.038. Epub 2016 Aug 29. PMID 27595443

RESULTS

PARTICIPANT FLOW:
Groups:
- CSL's IVV: Participants received a dose of the 2008 or 2009 Southern Hemisphere formulation of CSL's IVV
- Placebo: Participants received a dose of placebo in either 2008 or 2009 Southern Hemisphere influenza season
Period: Overall Study
Arm/Group | CSL's IVV | Placebo
Started | 10033 | 5011
Completed | 9827 | 4907
Not Completed | 206 | 104
Not completed — Adverse Event | 6 | 1
Not completed — Protocol Violation | 11 | 2
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Moved away from the study area | 20 | 9
Not completed — Lost to Follow-up | 132 | 71
Not completed — Reason not provided or not specified | 25 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSL's IVV | Placebo | Total
Number analyzed (Participants) | 10033 | 5011 | 15044
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10033 | 5011 | 15044
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (14.69) | 35.4 (14.69) | 35.5 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5523 | 2667 | 8190
  Male | 4510 | 2344 | 6854
Region of Enrollment [Number; unit: participants]
  Australia | 8201 | 4090 | 12291
  New Zealand | 1832 | 921 | 2753

OUTCOME MEASURES:

1. Primary Outcome: CSL's IVV Overall Vaccine Efficacy (VE) Versus Placebo Through Assessment of Incidence of Laboratory Confirmed Influenza A/B Infection
Description: Incidence of Laboratory Confirmed Influenza A/B infection was assessed per the study population in the 2008 and 2009 Southern Hemisphere influenza seasons.
  Vaccine efficacy = 100 x (1 - ratio of incidence rate). Ratio of incidence rate = active Study Vaccine recipient infection rate / placebo recipient infection rate.
Time Frame: 2008 and 2009 Southern Hemisphere influenza seasons, until 30 November 2009
Population: Evaluable Population for the Clinical Endpoint Analysis consisted of all participants who: received study vaccine and clinical endpoint follow-up was longer than 14 days after vaccination; and had not taken any contraindicated medications during the On-study or Clinical Endpoint Periods as potentially impacting clinical endpoint assessments.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 9889 | 4960
Ratio | 2.24 [1.97 to 2.57] | 3.87 [3.37 to 4.44]
Statistical Analysis 1: Comparison: CSL's IVV vs Placebo; Vaccine efficacy = 100 x (1 - ratio of incidence rate); Test type: Superiority or Other; Vaccine Efficacy = 42, 95% CI 2-sided [30 to 52]

2. Secondary Outcome: CSL's IVV Vaccine Efficacy Versus Placebo Through Assessment of Incidence of Laboratory Confirmed Influenza A/B Infection Due to Strains Matched to Vaccine Strains
Description: Incidence of laboratory confirmed influenza A/B infection due to strains matched to vaccine strains was assessed per the study population in the 2008 and 2009 Southern Hemisphere influenza seasons.
  Vaccine efficacy = 100 x (1 - ratio of incidence rate). Ratio of incidence rate = active Study Vaccine recipient infection rate / Placebo recipient infection rate.
Time Frame: 2008 and 2009 Southern Hemisphere influenza seasons, until 30 November 2009
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 9889 | 4960
Ratio | 0.59 [0.45 to 0.76] | 1.47 [1.17 to 1.85]
Statistical Analysis 1: Comparison: CSL's IVV vs Placebo; Vaccine efficacy = 100 x (1 - ratio of incidence rate); Test type: Superiority or Other; Vaccine efficacy = 60, 95% CI 2-sided [44 to 72]

3. Secondary Outcome: Incidence of Influenza-like Illness (ILI)
Description: The criteria for the protocol defined ILI were as follows:
  * At least one respiratory symptom:
  * cough, sore throat or nasal congestion
  * And at least one systemic symptom:
  * fever (as defined by oral temperature ≥ 37.8°C (100.0°F), or feverishness (as defined by participant's subjective feeling of fever), chills or body aches.
  The CDC ILI case definition was the occurrence of fever (100°F [37.8°C] or higher) in conjunction with either cough or sore throat.
Time Frame: 2008 and 2009 Southern Hemisphere influenza seasons, until 30 November 2009
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 9889 | 4960
Percentage of participants
  Reported ILI (protocol definition) | 11.9 | 13.5
  Culture-confirmed ILI | 1.5 | 2.4
  Reported ILI (CDC definition) | 2.6 | 3.6
  Laboratory-confirmed ILI (CDC definition) | 0.9 | 1.7

4. Secondary Outcome: Percentage of Participants With a Minimum Post-vaccination Hemagglutination Inhibition (HI) Titer of 1:40, Year 2008
Time Frame: 21 days after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 303 | 147
Percentage of participants
  H1N1 (A/Solomon Islands/3/2006) | 99 [97 to 100] | 42 [34 to 51]
  H3N2 (A/Brisbane/10/2007) | 97 [94 to 98] | 35 [27 to 43]
  B (B/Brisbane/3/2007) | 77 [72 to 82] | 13 [8 to 19]

5. Secondary Outcome: Percentage of Participants With a Minimum Post-vaccination Hemagglutination Inhibition (HI) Titer of 1:40, Year 2009
Time Frame: 21 days after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 291 | 149
Percentage of participants
  H1N1 (A/Brisbane/59/2007) | 94 [90 to 96] | 36 [28 to 44]
  H3N2 (A/Uruguay/2007) | 94 [90 to 96] | 43 [35 to 51]
  B (B/Florida/4/2006) | 89 [85 to 93] | 30 [23 to 38]

6. Secondary Outcome: Percentage of Participants With Seroconversion 21 Days After Study Vaccination, Year 2008
Description: Seroconversion rate: defined as the percentage of participants with either a pre-vaccination HI titer < 1:10 and a post-vaccination HI titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and a minimum four-fold rise in post-vaccination HI antibody titer.
Time Frame: 21 days after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 303 | 147
Percentage of participants
  H1N1 (A/Solomon Islands/3/2006) | 81 [76 to 85] | 1 [0 to 4]
  H3N2 (A/Brisbane/10/2007) | 87 [82 to 90] | 1 [0 to 4]
  B (B/Brisbane/3/2007) | 63 [57 to 69] | 1 [0 to 4]

7. Secondary Outcome: Percentage of Participants With Seroconversion 21 Days After Study Vaccination, Year 2009
Description: as for outcome 6
Time Frame: 21 days after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 291 | 149
Percentage of participants
  H1N1 (A/Brisbane/59/2007) | 78 [72 to 82] | 1 [0 to 4]
  H3N2 (A/Uruguay/2007) | 81 [76 to 85] | 1 [0 to 5]
  B (B/Florida/4/2006) | 61 [55 to 67] | 0 [0 to 0]

8. Secondary Outcome: Geometric Mean Fold Increase in HI Titer 21 Days After Study Vaccination, Year 2008
Description: Geometric mean fold increase in HI titer was defined as the geometric mean titer (GMT) after vaccination divided by the GMT before vaccination.
Time Frame: 21 days after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Fold increase
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 303 | 147
Fold increase
  H1N1 (A/Solomon Islands/3/2006) | 21 [17 to 26] | 1 [1 to 1]
  H3N2 (A/Brisbane/10/2007) | 18 [15 to 21] | 1 [1 to 1]
  B (B/Brisbane/3/2007) | 8 [7 to 10] | 1 [1 to 1]

9. Secondary Outcome: Geometric Mean Fold Increase in HI Titer Rate 21 Days After Study Vaccination, Year 2009
Description: as for outcome 8
Time Frame: 21 days after study vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Fold increase
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 291 | 149
Fold increase
  H1N1 (A/Brisbane/59/2007) | 13 [11 to 16] | 1 [1 to 1]
  H3N2 (A/Uruguay/2007) | 15 [13 to 18] | 1 [1 to 1]
  B (B/Florida/4/2006) | 6 [5 to 7] | 1 [1 to 1]

10. Secondary Outcome: Frequency and Intensity of Local and Systemic Solicited Symptoms
Description: Adverse event grading:
  Grade 1 (mild): Symptoms were easily tolerated and did not interfere with daily activities.
  Grade 2 (moderate): Discomfort was enough to cause some interference with daily activities.
  Grade 3 (severe): Symptoms that prevented normal, everyday activities.
  Fever Grade 1: ≥ 37.7°C - < 38.0°C (≥ 99.9 - < 100.4°F) Grade 2: ≥ 38.0°C - < 39.0°C (≥ 100.4 - < 102.2°F) Grade 3: ≥ 39.0°C (> 102.2°F)
Time Frame: 5 days after study vaccination
Population: Safety Population comprised all participants who received study vaccine (CSL's IVV or placebo) and provided at least one safety assessment after the vaccination.
Measure: Number; unit: Participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 10015 | 5005
Participants
  Any local solicited symptom | 7474 | 1021
  Any pain | 4850 | 539
  Grade 3 pain | 19 | 0
  Any tenderness | 6956 | 874
  Grade 3 tenderness | 30 | 2
  Any redness | 362 | 18
  Grade 3 redness | 3 | 0
  Any swelling / induration | 433 | 20
  Grade 3 swelling / induration | 6 | 0
  Any bruising | 135 | 29
  Grade 3 bruising | 1 | 0
  Any systemic solicited symptom | 4670 | 1955
  Any fever | 258 | 93
  Grade 3 fever | 8 | 2
  Any headache | 2553 | 1176
  Grade 3 headache | 43 | 19
  Any malaise | 2916 | 1277
  Grade 3 malaise | 67 | 24
  Any myalgia | 2150 | 609
  Grade 3 myalgia | 33 | 5
  Any chills | 509 | 187
  Grade 3 chills | 17 | 3
  Any nausea | 678 | 287
  Grade 3 nausea | 22 | 16
  Any vomiting | 83 | 38
  Grade 3 vomiting | 10 | 4

11. Secondary Outcome: Frequency and Intensity of Unsolicited Adverse Events (UAEs)
Description: UAE grading:
  Grade 1 (mild): Symptoms were easily tolerated and did not interfere with daily activities.
  Grade 2 (moderate): Discomfort was enough to cause some interference with daily activities.
  Grade 3 (severe): Symptoms that prevented normal, everyday activities.
Time Frame: 21 days after study vaccination
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 9889 | 4960
Participants
  Number of participants with at least one UAE | 3519 | 1698
  Number of participants reported Grade 1 UAE | 1604 | 750
  Number of participants reported Grade 2 UAE | 1536 | 784
  Number of participants reported Grade 3 UAE | 378 | 162

12. Secondary Outcome: Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence that at any dose:
  * Resulted in death;
  * Was life-threatening;
  * Required an unexpected in-participant hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability / incapacity;
  * Was a congenital anomaly / birth defect; and / or
  * Was medically significant (defined as an event that did not necessarily meet any of the SAE criteria, but was judged by the treating physician to potentially jeopardize the participant or require medical intervention to prevent one of the out
Time Frame: 180 days after study vaccination
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 9889 | 4960
Participants
  Number of participants with at least one SAE | 100 | 44
  Number rof participants with related SAE | 0 | 0

13. Secondary Outcome: New Onsets of Chronic Illness (NOCI)
Description: An NOCI was defined as the diagnosis of a chronic medical condition where the symptoms commenced or worsened following exposure to study vaccine and may have included those potentially controllable by medication (e.g., glaucoma, hypertension).
Time Frame: 180 days after study vaccination
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | CSL's IVV | Placebo
Number analyzed (Participants) | 9889 | 4960
Participants
  Number of participants with at least one NOCI | 80 | 46
  Number of participants with related NOCI | 3 | 0

ADVERSE EVENTS:
Time Frame: 21 days after study vaccination for unsolicited adverse events and 180 days after study vaccination for serious adverse events.
Description: Other adverse events presented were unsolicited adverse events up to 21 days after study vaccination
Arm/Group | CSL's IVV | Placebo
Serious Adverse Events (participants affected / at risk) | 100/10015 | 44/5005
Other Adverse Events (participants affected / at risk) | 3028/10015 | 1549/5005
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL's IVV (N=10015) | Placebo (N=5005)
Appendicitis (Infections and infestations) | 8 (8) | 2 (2)
Cellulitis (Infections and infestations) | 4 (4) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Vestibular neuronitis (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Measles (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pyomyositis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Infections and infestations) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ruptured ectopic pregnancy (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (2)
Heart injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL's IVV (N=10015) | Placebo (N=5005)
Upper respiratory tract infection (Infections and infestations) | 387 (402) | 201 (205)
Headache (Nervous system disorders) | 1128 (1567) | 558 (712)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 501 (529) | 258 (276)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 248 (273) | 150 (160)
Cough (Respiratory, thoracic and mediastinal disorders) | 220 (228) | 104 (112)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 155 (163) | 80 (82)
Back pain (Musculoskeletal and connective tissue disorders) | 135 (155) | 70 (78)
Dysmenorrhea (Reproductive system and breast disorders) | 144 (148) | 73 (77)
Nasopharyngitis (Infections and infestations) | 110 (113) | 55 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less